CLINICAL TRIAL: NCT05210725
Title: Trained Immunity by Dual-pathway Inhibition (Low-dose Rivaroxaban and Acetylsalicylic Acid) in Coronary Artery Disease'
Brief Title: Trained Immunity by Dual-pathway Inhibition in Coronary Artery Disease
Acronym: DUALCAD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL2021-13291
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stable coronary artery disease (Experimental): Patients with stable coronary artery disease with an indication for single antiplatelet therapy according to international (ESC) guidelines, with a high cardiovascular risk.
  Interventions: Drug: Rivaroxaban 2.5 Mg Oral Tablet

INTERVENTIONS:
Drug: Rivaroxaban 2.5 Mg Oral Tablet — 2.5 mg rivaroxaban twice a day in addition to acetylsalicylic acid (80-00mg once a day, standard care).

SUMMARY:
Coronary artery disease (CAD) is a manifestation of systemic atherosclerosis for which single antiplatelet therapy (SAPT) is indicated if patients are stable. Recently dual pathway inhibition (DPI) by combining a low-dose factor Xa inhibitor (rivaroxaban2.5mg twice daily) with a single platelet inhibitor (ASA) has been demonstrated to be beneficial in treating CAD. The exact mechanisms underlying the benefits of DPI, are not completely understood. CAD is characterised by a state of chronic low-grade inflammation, where monocytes from CAD patients have a higher immune responsiveness to ex vivo stimulation with lipopolysaccharide (LPS) compared to healthy matched controls. Surprisingly, the investigators have recently observed an elevation in ex vivo immune responsiveness to LPS stimulation when switching from ASA monotherapy to DPI of ASA combined with rivaroxaban inpatients with peripheral arterial disease (n=11; unpublished). Remarkably this was associated with no changes in systemic inflammation, as determined by Olink proteomics analysis. These findings suggest that factor Xa inhibitors can enhance immune cell responsiveness despite being clinically beneficial to CAD. The exact mechanisms contributing to the observed increased immune responsiveness remain unexplored.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* stable CAD
* with an indication for single antiplatelet therapy according to international (ESC) guidelines,
* high cardiovascular risk based on a SMART risk score [9] of at least 20% and/or the judgement of the cardiologist
* at least 1 year after myocardial infarction or multivessel CAD
* >16 years old
* Written informed consent

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Use of more intensive antithrombotic treatment (dual antiplatelet therapy, DPI, direct oral anticoagulants, vitamin k antagonists)
* Use of immunosuppressant and/or anti-inflammatory therapy, including glucocorticoids, cytostatics, antibodies, immunophilins, interferons, Tumor Necrosis Factor (TNF) binding proteins, mycophenolate and interleukin antagonists
* Contra-indication to rivaroxaban

  * Hypersensitivity to rivaroxaban
  * at significant risk for major bleeding

    * current gastrointestinal ulceration
    * presence of malignant neoplasms, with the exception of non-melanoma skin cancer
    * recent (<2 months) brain or spinal injury
    * recent (<3 months) brain or spinal surgery
    * recent (<3 months) intracranial, gastrointestinal or pulmonary hemorrhage
    * presence of arteriovenous malformations,
    * major intraspinal or intracerebral vascular abnormalities
    * congenital or acquired bleeding disorders
    * uncontrolled severe arterial hypertension (180 mmHg or more systolic, or 110 mmHg or more diastolic)
  * Severe hepatic disease: Child Pugh B or C [10]
  * Severe kidney failure: estimated glomerular filtration rate<15 ml/min or requiring dialysis
  * severe heart failure with known ejection fraction < 30% or New York Heart Association class III or IV symptoms [12]
  * concomitant treatment with medication with a strong pharmacokinetic interaction with rivaroxaban, leading to contra-indication according to the "regionale_NOAC_richtlijn" [12]
* Pregnant or breastfeeding women
* Unable to give informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Whole blood immune responsiveness | 12 weeks
  Change in whole blood immune responsiveness to lipopolysaccharide stimulation when switching from acetylsalicylic acid to dual pathway inhibition (acetylsalicylic acid and low-dose rivaroxaban).

SECONDARY OUTCOMES:
White blood cell count and distribution | 3 months
  changes in white blood cell count and distribution when switching from acetylsalicylic acid to dual pathway inhibition (acetylsalicylic acid and low-dose rivaroxaban).
Monocyte immune responsiveness | 3 months
  Change in monocyte immune responsiveness to LPS stimulation when switching from acetylsalicylic acid to dual pathway inhibition (acetylsalicylic acid and low-dose rivaroxaban).
Enrichment of epigenetic marks on genes | 3 months
  Enrichment of epigenetic marks on genes when switching from acetylsalicylic acid to dual pathway inhibition (acetylsalicylic acid and low-dose rivaroxaban).

CONTACTS AND LOCATIONS:
Overall Officials: Saloua El Messaoudi, MD PhD, Study Director — Radboud University Medical Center; Michiel C Warlé, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Groh LA, Willems LH, Fintelman P, Reijnen MMPJ, El Messaoudi S, Warle MC. Dual-Pathway Inhibition with Rivaroxaban and Low-Dose Aspirin Does Not Alter Immune Cell Responsiveness and Distribution in Patients with Coronary Artery Disease. Cardiol Ther. 2024 Mar;13(1):233-242. doi: 10.1007/s40119-023-00342-5. Epub 2023 Dec 6. PMID 38055176